CLINICAL TRIAL: NCT02619799
Title: A Comparative Study Between Intrathecal Magnesium Sulphate Versus Midazolam Along With Epidural 0.75% Ropivacaine in Combined Spinal Epidural Technique for Preeclampsia Parturients Undergiong Elective Caesarean Section
Brief Title: A Comparative Study of Intrathecal Magnesium Sulphate & Midazolam With Epidural Ropivacaine for Caesarean Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rangaraya Medical College (Other)
Responsible Party: Principal Investigator, Dr. Paleti Sophia, Principle investigator, Rangaraya Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rangaraya medical college
Record Dates: First submitted 2015-11-19; First posted 2015-12-02 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Pain
Keywords: magnesium sulphate; intrathecal route; midazolam
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP A(MAGNESIUM GROUP) (Active Comparator): MAGNESIUM GROUP received 50 mg(0.1 ml) of intrathecal magnesium sulphate diluted to 1 ml with 0.9% normal saline combined with 14-16 ml of epidural 0.75% ropivacaine as a part of combined spinal epidural technique at L2-L3/L3-L4 interspace.
  Interventions: Drug: intrathecal magnesium sulphate,
- GROUP B(MIDAZOLAM GROUP) (Active Comparator): MIDAZOLAM GROUP received 1mg(0.2ml) of intrathecal midazolam diluted to 1ml with 0.9% normal saline combined with 14-16 ml of epidural 0.75% ropivacaine as a part of combined spinal epidural technique at L2-L3/L3-L4 interspace.
  Interventions: Drug: Intrathecal midazolam

INTERVENTIONS:
Drug: intrathecal magnesium sulphate, — comparision of effects of intrathecal magnesium sulphate with intrathecal midazolam when administered along with epidural 0.75% Ropivacaine
  Other Names: Magneon
  Arms: GROUP A(MAGNESIUM GROUP)
Drug: Intrathecal midazolam — comparision of effects of intrathecal magnesium sulphate with intrathecal midazolam when administered along with epidural 0.75% Ropivacaine
  Other Names: Mizolam
  Arms: GROUP B(MIDAZOLAM GROUP)

SUMMARY:
This study compares whether addition of Magnesium or Midazolam intrathecally to epidurally administered isobaric Ropivacaine improves the quality of blockade, haemodynamics and duration of analgesia post-operatively. 25 parturients were given intrathecal Magnesium and rest of the 25 parturients were given intrathecal Midazolam combined with 0.75% Ropivacaine via epidural route.

DETAILED DESCRIPTION:
Magnesium sulphate and Midazolam have been used in clinical trials as adjuvants to local anaesthetics via intrathecal and epidural routes and are effective in augmenting the quality of block and prolonging post-operative analgesia.

Noxious stimulation leads to the release of glutamate and aspartate neuratransmitters which bind to various sub-classes of excitatory aminoacid, including the NMDA receptor. Intrathecal magnesium potentiates neuraxial anaesthesia by blocking NMDA receptors with out causing significant side effects as reported in various studies.

Intrathecal Midazolam produces antinociception at spinal cord-level through benzodiazepine GABA-A receptor complex which are present abundantly in the lamina 2 of spinal cord. Midazolam also releases endogenous opioid acting at spinal delta receptors and also enhances adenosine release which also augments analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 50 pregnant women
* ASA-I and II parturients
* Weight 50-80 kgs
* Pre-eclampsia

Exclusion Criteria:

* Thrombocytopenia
* HELLP syndrome
* Parturients on magnesium therapy
* Foetal distress
* Parturients on benzodiazepine therapy
* Patient refusal
* Contraindications to regional anaesthesia

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Culebras X, Gaggero G, Zatloukal J, Kern C, Marti RA. Advantages of intrathecal nalbuphine, compared with intrathecal morphine, after cesarean delivery: an evaluation of postoperative analgesia and adverse effects. Anesth Analg. 2000 Sep;91(3):601-5. doi: 10.1097/00000539-200009000-00019. PMID 10960384

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants] — parturients aged between 18-28 years were included in the study
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 25 | 25 | 50
    >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — female parturients who completed 37 weeks of gestational age and who are preeclamptic were included in the study
  participants
    female pregnant patients | 25 | 25 | 50
weight in kilograms [Mean (Standard Deviation); unit: kilograms] — parturients weighing between 50 -80 kilograms were included in the study
  kilograms | 68 (5) | 72 (6) | 70 (5.5)
age in years [Mean (Standard Deviation); unit: years] | 23 (2) | 26 (3) | 24.5 (2.5)
height in centimeters [Mean (Standard Deviation); unit: centimeters] — Parturients with height range between 150-170 cms were included in the study
  centimeters | 156 (3) | 158 (6) | 157 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Postoperative Analgesia
Description: pain is assessed using visual analogue scale every hour after completion of surgery until first 12 postoperative hours.
Time Frame: first 12 hours after completion of surgery.
Measure: Mean (Standard Deviation); unit: time in minutes
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP)
Number analyzed (Participants) | 25 | 25
time in minutes | 334 (39) | 280 (23.4)

2. Secondary Outcome: Onset of Sensory Blockade
Description: the onset time of sensory blockade was assessed with pinprick .
Time Frame: every 2- 3 minutes for initial 20 minutes ,then every 30 min intervals for first 6 -8 hrs after completion of surgery..
Measure: Mean (Standard Deviation); unit: time in minutes
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP)
Number analyzed (Participants) | 25 | 25
time in minutes | 9.86 (1.37) | 7.93 (0.87)

3. Secondary Outcome: Duration of Sensory Blockade
Description: the duration of sensory blockade was assessed with pinprick .
Time Frame: every 2- 3 minutes for initial 20 minutes ,then every 30 min intervals for first 6 -8 hrs after completion of surgery..
Measure: Mean (Standard Deviation); unit: time in minutes
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP)
Number analyzed (Participants) | 25 | 25
time in minutes | 295 (36) | 245 (26.4)

4. Secondary Outcome: Onset of Motor Blockade
Description: assessed with modified bromage scale.
Time Frame: every 5 minute intervals for initial 30 min , then every 30 minute intervals for first 6-8 hrs after completion of surgery.
Measure: Mean (Standard Deviation); unit: time in minutes
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP)
Number analyzed (Participants) | 25 | 25
time in minutes | 12.5 (1.6) | 7.68 (3.2)

5. Secondary Outcome: Duration of Motor Blockade
Description: assessed with modified bromage scale.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: time in minutes
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP)
Number analyzed (Participants) | 25 | 25
time in minutes | 265 (24.6) | 223 (22.2)

6. Secondary Outcome: Perioperative Side Effects
Description: through out the intraoperative period and initial 12 hours postoperatively parturients were assessed for PONV,sedation,respiratory depression hypotension ,bradycardia and shivering.
Time Frame: through out the intraoperative period and first 12 postoperative hours.
Measure: Number; unit: participants
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP)
Number analyzed (Participants) | 25 | 25
participants
  Nausea and vomiting | 2 | 3
  shivering | 1 | 3

ADVERSE EVENTS:
Time Frame: first 12 hours of postoperative period all the parturients were monitored for any adverse events like nausea,vomiting,shivering,respiratory depression and sedation.
Arm/Group | GROUP A(MAGNESIUM GROUP) | GROUP B(MIDAZOLAM GROUP)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GROUP A(MAGNESIUM GROUP) (N=25) | GROUP B(MIDAZOLAM GROUP) (N=25)
shivering (Surgical and medical procedures) | 1 (2) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes